CLINICAL TRIAL: NCT04965753
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Intravenously Administered FHD-609 in Subjects With Advanced Synovial Sarcoma or Advanced SMARCB1-Loss Tumors
Brief Title: FHD-609 in Subjects With Advanced Synovial Sarcoma or Advanced SMARCB1-Loss Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Foghorn Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHD-609-C-001
Record Dates: First submitted 2021-06-26; First posted 2021-07-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Advanced Synovial Sarcoma
Keywords: advanced synovial sarcoma; synovial sarcoma; SS; phase 1; FHD-609; BRD9; Foghorn; Foghorn Therapeutics; SMARCB1 loss; INI1 loss; poorly differentiated chordoma; epithelioid sarcoma; malignant rhabdoid tumor; SMARCB1; INI1
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma; Rhabdoid Tumor

STUDY DESIGN:
Intervention Model Description: Open label single arm dose escalation and three-arm expansion study in patients with advanced synovial sarcoma or advanced SMARCB1-loss tumors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FHD-609 (Experimental): Up to approximately 104 patients will be enrolled in dose escalation and expansion.
  Interventions: Drug: FHD-609

INTERVENTIONS:
Drug: FHD-609 — FHD-609 as a single, intravenously administered agent given twice-weekly (BIW). Alternative dosing regimens may be evaluated.

SUMMARY:
This Phase 1, multicenter, open-label, dose escalation and expansion study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of FHD-609 given intravenously in subjects with advanced synovial sarcoma or advanced SMARCB1-loss tumors.

DETAILED DESCRIPTION:
This study is an ascending multiple dose clinical trial with expansion arms. It is primarily intended to evaluate the safety and tolerability of FHD-609 when administered intravenously to subjects with advanced synovial sarcoma or advanced SMARCB1-loss tumors. The Dose Escalation Phase will allow for the determination of the recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) of FHD-609. This study will also evaluate the PK/PD profiles of multiple dose administration of FHD-609.

The Dose Expansion Phase will allow a more robust evaluation of the safety profile of FHD-609, including toxicities that may occur less frequently, and an assessment of anti-tumor activity. The data from this study in subjects with advanced synovial sarcoma, including safety, tolerability, PK/PD findings, and anti-tumor activity, will form the basis for subsequent clinical development of FHD-609.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 or ≥ 16 years of age with a minimum body weight of 50 kg.
2. Subject must have a diagnosis of SS or a SMARCB1-loss tumor:

   • SS:

   - Evidence of the SS18-SSX rearrangement and/or a confirmed pathologic diagnosis of SS must be available.

   May be treatment naïve or previously treated (see definition below)

   • SMARCB1-loss tumor:
   * A solid tumor primarily characterized by SMARCB1 loss (eg, malignant rhabdoid tumors, epithelioid sarcoma, poorly differentiated chordoma) Documentation of biallelic SMARCB1 alterations and/or corresponding protein loss, and/or a confirmed pathologic diagnosis of a solid tumor primarily characterized by SMARCB1 loss, must be available.
   * Other solid tumors with SMARCB1 loss. Documentation of biallelic SMARCB1 alterations and/or corresponding protein loss must be available.

   Note: Inclusion criterion 15 provides timing requirements for prior therapy.
3. Subject must have measurable disease by RECIST v1.1, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as ≥ 10 mm with calipers and/or CT scan. Measurable lesions cannot have undergone any local treatment or radiation unless the lesion has progressed post treatment nor can any local treatment or radiation involving measurable lesions be anticipated. Exceptions to the requirements for measurable disease may be made in discussion with the sponsor.
4. Subject or his/her parent or legal guardian (when applicable) must be able to understand and be willing to sign an informed consent and, when applicable, subject must sign assent form.
5. Subject must be willing and able to comply with scheduled study visits and treatment plans.
6. Subject must be willing to undergo all study procedures (biopsies at baseline, at least 1 on-treatment and at EOT [unless contraindicated due to medical risk; other exceptions to this are at the discretion of the Sponsor]), laboratory testing, and imaging approximately every 8 (or 12) weeks independent of dose delays, interruptions, and/or reductions.
7. Subject must have an ECOG PS of ≤ 2.

   • Arm 2 (Dose Expansion Phase): Subject must have an ECOG PS of ≤ 3
8. Subject must have a life expectancy of ≥ 3 months.

   • Arm 2 (Dose Expansion Phase): Subject must have a life expectancy of ≥ 2 months
9. Subject must have adequate venous access for IV drug administration and blood collection.
10. Subject must have adequate cardiac function as evidenced by:

    * LVEF of ≥ 40% by ECHO. Other methods of evaluating LVEF may be performed according to institutional practice.
    * Corrected QT interval (QTc) using Fridericia's formula (QTcF) < 470 msec
11. Subject must have adequate hepatic function as evidenced by:

    * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (≤ 3.0 × ULN for subjects with Gilbert's syndrome)
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3.0 × ULN (≤ 5.0 × ULN if liver metastases are present)
    * Alkaline phosphatase (ALP) ≤ 3.0 × ULN (≤ 5.0 × ULN if liver metastases are present and/or known bone disease is present)
    * No known portal vein thrombosis
12. Subject must have adequate renal function as evidenced by:

    • Glomerular filtration rate (GFR) ≥ 50 mL/min (based on a contemporary, widely accepted, and clinically applicable equation that estimates glomerular filtration rate or a measure of glomerular filtration rate [e.g. Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)])
13. Subject must have adequate hematologic function as evidenced by:

    * Hemoglobin ≥ 8 g/dL (Red blood cell [RBC] transfusions to achieve this level will be permitted up to 7 days prior to start of study drug and complete blood count [CBC] criteria for eligibility are confirmed within 24 hours of first study dose.)
    * White blood cells (WBCs) ≥ 2.0 × 109/L
    * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L
    * Platelets > 50 × 109/L (Transfusions to achieve this level will be allowed up to 72 hours prior to start of study drug.)
14. Subject must have adequate coagulation function as evidenced by:

    • International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN and partial thromboplastin time (PTT) ≤ 1.5 × ULN if not receiving anticoagulation therapy.

    Note: For subjects on anticoagulants, exceptions to these parameters are allowed if they are within the intended or expected range for their therapeutic use. Participants must have no history of clinically significant active bleeding (within 14 days of first dose of study drug) or pathological condition that carries high risk of bleeding (for example, tumor involving major vessels or known esophageal varices).
15. Timing requirements with respect to prior therapy and surgery are as follows:

    * At least 2 weeks or at least 5 half-lives, whichever is shorter, must have elapsed since administration of the last dose of any prior anticancer therapy (including investigational agents).
    * Subjects must be recovered from any clinically relevant effects of major surgery, laparoscopic procedure, or significant traumatic injury. Note: Central line placement, subcutaneous port placement, core biopsy, fine needle aspiration, and bone marrow biopsy/aspiration are not considered major surgeries.
    * For subjects who have received radiation therapy within 2 weeks of study start, health status must have returned to pre-radiation therapy baseline, and/or be adequate for study start, in the opinion of the Investigator. Radiation therapy cannot involve target lesions unless approved by the Sponsor.
16. Clinically significant toxicity related to prior therapy must have returned to ≤ Grade 1 by CTCAE by approximately 14 days prior to study start. Exceptions include Grade 2 alopecia and other Grade 2 toxicities determined to be stable and irreversible by the Investigator, and other well-controlled/stable toxicities, with approval of the Sponsor.
17. Female subjects must be:

    * Postmenopausal, defined as at least 12 months post-cessation of menses (without an alternative medical cause); or
    * Permanently sterile following documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or tubal ligation or having a male partner with vasectomy or having a female partner as affirmed by the subject; or
    * Nonpregnant, non-breastfeeding, and if sexually active having agreed to use a highly effective method of contraception (ie, hormonal contraceptives associated with inhibition of ovulation or intrauterine device [IUD], or intrauterine hormone-releasing system [IUS], or sexual abstinence) from Screening Visit until 187 days after final dose of study drug.
18. Male subjects must have documented vasectomy or if sexually active must agree to use a highly effective method of contraception with their partners of childbearing potential (ie, hormonal contraceptives associated with the inhibition of ovulation or IUD, or IUS, or sexual abstinence) from Screening until 97 days after final dose of study drug. Male subjects must agree to refrain from donating sperm during this time period.

Exclusion Criteria:

1. Subject (or parent or legal guardian, when applicable) is unable to provide informed consent (or assent, when applicable) and/or to follow protocol requirements.
2. Subject has other malignancy which may interfere with the diagnosis and/or treatment of SS/SMARCB1-loss tumors and/or interpretation of outcome results.
3. Subject has an active severe infection requiring systemic therapy. Subject is permitted to enroll once any required antibiotic and/or antifungal therapy has been completed and/or infection is determined to be controlled.
4. Subject has active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections; subjects with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Subject has known positive human immunodeficiency virus (HIV) antibody results or acquired immunodeficiency syndrome (AIDS)-related illness; subjects with CD4+ T-cell counts ≥ 350 cells/µL will be permitted, as will subjects who have not had an AIDS-related illness within the past 12 months.
5. Subject has an uncontrolled concurrent medical disease and/or psychiatric illness/social situation that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol.
6. Subject is requiring clinically significant or increasing doses of systemic steroid therapy for acute illness (stable doses for controlled chronic disease or symptoms are permitted) or any other systemic immunosuppressive medication. Stable doses of systemic immunosuppressive medications may be allowed with Sponsor approval. Local or targeted steroid and immunosuppressive therapies (eg, inhaled or topical steroids) are acceptable. See Exclusion criterion 7 for details on steroids in the setting of central nervous system (CNS) disease.
7. Subjects with known CNS metastases are only permitted under the following conditions: Brain metastases must have been stable for approximately 2 months since completion of most recent CNS-directed intervention. Subject may be receiving corticosteroids so long as the dose is stable or decreasing at the time of study entry. Anti-epileptic therapy is allowed so long as medications are not otherwise excluded and seizures have been controlled for approximately 4 weeks since the last anti-epileptic medication adjustment. Subjects with active brain metastases and/or leptomeningeal disease are excluded. Exceptions to this may be made on a case-by-case basis with approval of Sponsor.

   * Dose Escalation Phase: Subjects with known CNS metastases that meet the above conditions are permitted to enroll in dose escalation.
   * Arm 1 and Arm 3 (Dose Expansion Phase): Subjects with known or suspected CNS metastases are excluded from Arm 1 and Arm 3.
   * Arm 2 (Dose Expansion Phase): Subjects with CNS metastases that meet the above conditions are permitted to enroll in Arm 2.
8. Subject has known hypersensitivities to components of FHD-609.
9. Subject has prior exposure to a BRD9 degrader.
10. Subject is participating in any other clinical trials. Exceptions include participation in any observational or nontherapeutic clinical trials.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 31 months
  Dose escalation and expansion
Incidence of adverse events (AEs), serious adverse events (SAEs) including changes in safety laboratory parameters and AEs leading to discontinuation | Up to 31 months
  Dose escalation and expansion
Incidence of dose limiting toxicities (DLTs) | 6 weeks
  During first 6 weeks of treatment for each patient in dose escalation

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 30 months
  ORR is defined as the percentage of subjects achieving a complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Duration of Response (DOR) | Up to approximately 30 months
  DOR is defined as the time from first documented evidence of CR or PR until the earliest date of documented radiological progression per RECIST 1.1. or death due to any cause among subjects who achieved a CR or PR
Progression Free Survival (PFS) | Up to approximately 42 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression per RECIST 1.1. or death due to any cause, whichever happens first
Time to Response (TTR) | Up to approximately 30 months
  TTR is defined as the period of time from the date of first study drug administration until the first objective documentation of response per RECIST 1.1.
Overall Survival (OS) | Up to approximately 54 months
  OS is defined as the time from first dose of study treatment to the date of death, irrespective of the cause of death.
Plasma concentration of FHD-609 to characterize the pharmacokinetics (PK) parameters of FHD-609 | At multiple time points up to 6 weeks
  Plasma concentration of FHD-609 at the scheduled timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Reilly, MD, Study Director — Foghorn Therapeutics
Locations (12):
- United States (8):
  - City of Hope, Duarte, California
  - University of Miami Health System, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Istituto Nazionale dei Tumori, Milan, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Livingston JA, Blay JY, Trent J, Valverde C, Agulnik M, Gounder M, Le Cesne A, McKean M, Wagner MJ, Stacchiotti S, Agresta S, Quintas-Cardama A, Reilly SA, Healy K, Hickman D, Zhao T, Ballesteros-Perez A, Khalil A, Collins MP, Piel J, Horrigan K, Lefkovith A, Innis S, Lazar AJ, Cote GM, Wagner AJ. A Phase I Study of FHD-609, a Heterobifunctional Degrader of Bromodomain-Containing Protein 9, in Patients with Advanced Synovial Sarcoma or SMARCB1-Deficient Tumors. Clin Cancer Res. 2025 Feb 17;31(4):628-638. doi: 10.1158/1078-0432.CCR-24-2583. PMID 39660994